CLINICAL TRIAL: NCT05408546
Title: Evaluation of the Safety and Thrombolytic Effects of Ascending Doses of TS23 in Subjects With Intermediate-Risk (Sub-Massive) Acute Pulmonary Embolism
Brief Title: Novel α2-Antiplasmin Inactivation for Lysis of Intravascular Thrombi (NAIL-IT) Trial
Acronym: NAIL-IT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Translational Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TS23-U201
Record Dates: First submitted 2022-05-21; First posted 2022-06-07 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo + standard of care (SOC) anticoagulation
  Interventions: Drug: Placebo
- Low dose TS23 (Experimental): TS23 low dose + SOC anticoagulation
  Interventions: Drug: TS23
- Intermediate dose TS23 (Experimental): TS23 medium dose + SOC anticoagulation
  Interventions: Drug: TS23
- Higher dose TS23 (Experimental): TS23 highest dose + SOC anticoagulation
  Interventions: Drug: TS23

INTERVENTIONS:
Drug: TS23 — Monoclonal antibody to a2-antiplasmin
  Arms: Higher dose TS23; Intermediate dose TS23; Low dose TS23
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Phase II trial of TS23

DETAILED DESCRIPTION:
Evaluation of safety and thrombolytic effect of ascending doses of TS23 in subjects with intermediate-risk (sub-massive) acute pulmonary embolism (PE)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, age >18 years;
2. PE involving a segmental or more proximal pulmonary artery confirmed by CTPA scan and with an onset of symptoms not more than 5 days prior to diagnosis;
3. Subject is hemodynamically stable with a systolic blood pressure (SBP) >90 mm Hg;
4. Subject has evidence of RV dysfunction as indicated by a right ventricular-to-left ventricular (RV/LV) diameter ratio > 0.9 on CTPA scan (measuring the minor axis of the right and left ventricle in the transverse plane), prior to the initiation of study drug administration.

Exclusion Criteria:

1. Subjects for whom thrombolytic therapy or thrombectomy is planned; or subjects with history of administration of thrombolytic agents within the previous 4 days;
2. Subjects receiving ≥ 48 hours of therapeutic doses of heparin or low molecular weight heparin (LMWH) or other anticoagulant therapy immediately prior to randomization;
3. Subjects with contraindications to SOC therapies such as unfractionated heparin or LMWH or oral anticoagulant, or any of the excipients (including study drug excipients);
4. Subjects who are considered at very high risk of bleeding:

   1. Known coagulation disorder with history of pathologic bleeding tendencies
   2. Subjects with prior intracranial hemorrhage, known arteriovenous malformation or aneurysm of the brain, or evidence of active bleeding;
   3. Subjects with a history of major surgery, clinically significant head trauma (in the opinion of the Principal Investigator), or stroke in the past 3 months prior to randomization;
   4. Subjects with uncontrolled hypertension defined as SBP ≥180 mm Hg and/or diastolic BP (DBP)

      ≥110 mm Hg at randomization
   5. Subjects requiring concomitant dual antiplatelet therapy
5. Subjects with Creatinine Clearance (CrCL) < 30 mL/min or serum creatinine ≥ 2.5 mg/dL;
6. Subjects with hemoglobin < 8.0 g/dL;
7. Subjects with a platelet count < 100,000/µL;
8. Subjects with acute or persistent hepatitis or diagnosed active liver disease or with elevation of liver enzymes: Alanine transaminase (ALT) or aspartate transaminase (AST) ≥ 3 x upper limit of normal (ULN);
9. Subjects with known history of testing positive for Hepatitis B antigen or Hepatitis C antibody;
10. Subjects with known history of testing positive for the human immunodeficiency virus (HIV);
11. Subjects with life-expectancy < 6 months;
12. Female subjects of child bearing potential with a positive pregnancy test or who are lactating, or unwilling to use highly effective methods of contraception. Highly effective methods of birth control include combination hormonal therapy (estrogen and progresterone), contraceptives administered orally, intravaginally or transdermally, progesterone-only contraceptives administered orally, by injection or implantation, use of an intrauterine device (IUD), intrauterine hormone- releasing system (IUS), bilateral tubal occlusion, partner vasectomy or sexual abstinence;
13. Subjects currently participating in another investigational study or who have participated in an investigational drug study within 30 days (or longer depending on the half-life of the investigational drug; should allow at least five half-life of the investigational drug) prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
RV/LV | 48 hours after treatment
  Ratio of the right to left ventricle dimensions on CT perfusion angiogram (CTPA)
Safety- Bleeding | within 7 days of treatment
  Frequency of major or clinically significant bleeding

SECONDARY OUTCOMES:
Thrombus dissolution | 48 hours after treatment
  Change in modified Miller Score

CONTACTS AND LOCATIONS:
Overall Officials: Guy L Reed, MD, Principal Investigator — Translational Sciences
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh S, Houng A, Reed GL. Releasing the Brakes on the Fibrinolytic System in Pulmonary Emboli: Unique Effects of Plasminogen Activation and alpha2-Antiplasmin Inactivation. Circulation. 2017 Mar 14;135(11):1011-1020. doi: 10.1161/CIRCULATIONAHA.116.024421. Epub 2016 Dec 27. PMID 28028005
- [Background] Singh S, Houng AK, Reed GL. Venous stasis-induced fibrinolysis prevents thrombosis in mice: role of alpha2-antiplasmin. Blood. 2019 Sep 19;134(12):970-978. doi: 10.1182/blood.2019000049. Epub 2019 Aug 8. PMID 31395599
- [Background] Reed GL, Houng AK, Wang D. Microvascular thrombosis, fibrinolysis, ischemic injury, and death after cerebral thromboembolism are affected by levels of circulating alpha2-antiplasmin. Arterioscler Thromb Vasc Biol. 2014 Dec;34(12):2586-93. doi: 10.1161/ATVBAHA.114.304530. Epub 2014 Sep 25. PMID 25256235
- [Background] Houng AK, Wang D, Reed GL. Reversing the deleterious effects of alpha2-antiplasmin on tissue plasminogen activator therapy improves outcomes in experimental ischemic stroke. Exp Neurol. 2014 May;255:56-62. doi: 10.1016/j.expneurol.2014.02.009. Epub 2014 Feb 18. PMID 24556477
- [Background] Cesarman-Maus G, Hajjar KA. Molecular mechanisms of fibrinolysis. Br J Haematol. 2005 May;129(3):307-21. doi: 10.1111/j.1365-2141.2005.05444.x. PMID 15842654
- [Background] Meyer G, Vicaut E, Konstantinides SV. Fibrinolysis for intermediate-risk pulmonary embolism. N Engl J Med. 2014 Aug 7;371(6):581-2. doi: 10.1056/NEJMc1406283. No abstract available. PMID 25099590
- [Background] Aghayev A, Furlan A, Patil A, Gumus S, Jeon KN, Park B, Bae KT. The rate of resolution of clot burden measured by pulmonary CT angiography in patients with acute pulmonary embolism. AJR Am J Roentgenol. 2013 Apr;200(4):791-7. doi: 10.2214/AJR.12.8624. PMID 23521450
- [Background] Meinel FG, Nance JW Jr, Schoepf UJ, Hoffmann VS, Thierfelder KM, Costello P, Goldhaber SZ, Bamberg F. Predictive Value of Computed Tomography in Acute Pulmonary Embolism: Systematic Review and Meta-analysis. Am J Med. 2015 Jul;128(7):747-59.e2. doi: 10.1016/j.amjmed.2015.01.023. Epub 2015 Feb 11. PMID 25680885
- [Background] Ouriel K, Ouriel RL, Lim YJ, Piazza G, Goldhaber SZ. Computed tomography angiography with pulmonary artery thrombus burden and right-to-left ventricular diameter ratio after pulmonary embolism. Vascular. 2017 Feb;25(1):54-62. doi: 10.1177/1708538116645056. Epub 2016 Jul 9. PMID 27090586
- [Background] Zuo Z, Yue J, Dong BR, Wu T, Liu GJ, Hao Q. Thrombolytic therapy for pulmonary embolism. Cochrane Database Syst Rev. 2021 Apr 15;4(4):CD004437. doi: 10.1002/14651858.CD004437.pub6. PMID 33857326